CLINICAL TRIAL: NCT04638530
Title: Breaking Bad News to Family Members in a Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Linda R Duska, professor of obstetrics and gynecology and associate dean for clinical research at UVA School of Medicine., University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3977
Record Dates: First submitted 2020-10-11; First posted 2020-11-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Resident Education, Patient Communication, Breaking Bad News to Patients Remotely, Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residents (Other): All residents will participate in the activity
  Interventions: Other: Education on breaking bad news to family members remotely

INTERVENTIONS:
Other: Education on breaking bad news to family members remotely — Participants will receive a combination of surveys, pre- and post-tests, lectures and didactics to increase their awareness of techniques to communicate difficult topics with patients remotely as well as skill building exercises.

SUMMARY:
Resident education on breaking bad news and conducting end of life conversations has been shown to improve comfort levels with having these conversations. Interventions with OB/GYN residents specifically have used a combination of didactics, resident role-playing and ultimately interaction with standardized patients with feedback from palliative care specialists. These interventions can be costly and also are not practical during the pandemic training environment where resident has transitioned to a virtual curriculum. While the didactics portions of this previously proven curriculum can be done virtually, the standardized patient interactions are challenging to replicate. Additionally, one of the key changes to patient care that has emerged during the pandemic is restrictive hospital and clinic visitor policies. Care providers must now have the ability to have difficult conversations and break bad news to family members over the phone rather than in person. Additionally, there has been an increasing reliance on telehealth visits. There are no currently studied training interventions in obstetrics and gynecology that address these skills.

DETAILED DESCRIPTION:
First residents will be asked to participate. After giving consent, they will complete a pre-study questionnaire regarding their education and experience with end of life and breaking bad news conversations: They will be queried on basic demographic information: Age, Sex, Year of Residency, Intended specialty, prior education on end of life and breaking bad news: (0 hrs, 1-3 hours, 4-10 hours, 10-40 hrs, > 40 hrs), prior palliative or hospice rotation, have you had interaction with palliative care providers during training, have you experienced the death of a close family member or friend?, have you experienced a personally life threatening diagnosis?. We also will query the number of times residents have participated in code discussions, breaking bad news, discussion about prognosis, discussion about care at the end of life and discussion about hospice. They will also rate their own ability and comfort with the following topics : self-assessed preparation and attitudes about end-of life communication. First will be asked to review "Discussing Resuscitation Preferences with Patients: Challenges and Rewards" There will be a didactic session during which we will review the article and discuss strategies for breaking bad news to family members. A faculty member from General OB/GYN, MFM and Gynecologic Oncology will each give a brief 10 min lecture on how they have difficulty conversations with patients and family members in their specific field (post-operative complications , pre-viable delivery, and hospice/end of life/withdrawal of car). The lecture will be taped for those unable to attend. Two sessions will be held during didactics via Zoom in two different months to encompass those on night shifts and vacations. Residents will be split into groups of 3 with a faculty member in each group. They will role-play three scenarios one specific to each of the subspecialties- 1) Pre-viable delivery, 2) Discussion of withdrawal of care for a patient with advanced gynecologic malignancy who can no longer make their own medical decisions, and 3) Telling a family member about a surgical complication requiring an emergent return to the operating room. One resident will play the part of the family member receiving the phone call. To better mimic phone conversation, video will be turned off during this portion. The faculty member will score the interaction based on the following criteria and also give specific feedback regarding what went well and what should be improved. After receiving feedback from the role playing session, residents will then sign up for a recorded session with an actor playing a family member. They will be randomly assigned to one of the three topics and will then be assessed by a faculty member with the same criteria. After each of the three sections of teaching, residents will be asked to rate on a 1 to 5 scale their experience with the content and if it improved their ability to have end of life conversations. 3 months following the intervention, residents will be queried with the same questions asked previously to assess changes in their comfort with these conversations

ELIGIBILITY:
Inclusion Criteria:

* residents in University of Virginia's residency in Obstetrics and Gynecology
* able to provide informed consent

Exclusion Criteria:

* under age 18
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pre vs. post test scores | 4 years
  Increase in self-reported comfort levels post education sessions compared to the "Bad News" pre-test questionnaire with ranking comfort level for a variety of breaking bad news scenarios from 1 to 5 with 5 indicating very comfortable and 1 indicating very uncomfortable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No